CLINICAL TRIAL: NCT02522650
Title: A Crossover Pilot Study of the Effect of Amiloride on Proteinuria in Patients With Proteinuric Kidney Disease
Brief Title: A Crossover Pilot Study of the Effect of Amiloride on Proteinuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Wen Shen, MD, PHD, Associate Professor of Medicine, Georgetown University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0496
Record Dates: First submitted 2015-07-23; First posted 2015-08-13 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Proteinuria
Keywords: amiloride; proteinuric kidney disease; urokinase plasminogen activator receptor; proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Amiloride; Triamterene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amiloride Phase (Experimental): Subject receives 5mg of Amiloride twice daily for 8 weeks.
  Interventions: Drug: Amiloride
- Triamterene Phase (Active Comparator): Subject receives 50mg of Triamterene twice daily for 8 weeks.
  Interventions: Drug: Triamterene
- Washout Phase (No Intervention): Subject does not take any study medication for 4 weeks

INTERVENTIONS:
Drug: Amiloride — 5mg twice a day for 8 weeks
  Arms: Amiloride Phase
Drug: Triamterene — 50mg twice a day for 8 weeks
  Arms: Triamterene Phase

SUMMARY:
This cross-over study is designed to test the hypothesis that amiloride will reduce urinary protein excretion and protect the kidney from rapid progression in proteinuric kidney disease.

DETAILED DESCRIPTION:
Patients with proteinuric kidney disease will be enrolled and receive either amiloride or triamterene first, a similar diuretic acting on epithelial sodium channel (ENaC) as amiloride, but not inhibiting urokinase plasminogen activator receptor (uPAR), will be used as a control. Then patients will cross over to receive another medication. We postulate that amiloride could be beneficial in the patients with proteinuric kidney diseases and could be used as an adjunct therapy to reduce proteinuria and to delay renal disease progression in this patient population.

Specific Aim 1: To examine the effects of amiloride on 24 hour urine protein excretion in patients with proteinuric kidney diseases.

Specific Aim 2: To study if the effect of amiloride on proteinuria reduction is mediated by suppressing soluble urokinase plasminogen activator receptor (suPAR) expression.

Study Design:

The study includes 3 phases. 30 patients will be recruited to this study. All patients need to be on an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB) daily at least two month prior to the study.

Phase 1: Patients will be randomized to receive either amiloride 5mg twice daily or triamterene 50mg twice daily for 8 weeks. Serum potassium will be monitored one week before and one week after starting phase 1. If serum potassium remains equal to or less than 5.0mmol/L, amiloride or triamterene will be continued at same dose until the end of phase 1. If serum potassium is equal to or above 5.5 mmol/L, the patient will exit the study, and an adverse event will be reported. If serum potassium is between 5.1-5.4 mmol/L, it will be monitored again in one week. If serum potassium is above 5.5 mmol/L, the patient will exit the study, and an adverse event will be reported. If serum potassium remains in the same range, the patient will continue amiloride or triamterene at the same dose to complete phase 1.

Phase 2: the patients will discontinue amiloride or triamterene for a washout for 4 weeks, but continue with the ACE inhibitor or ARB.

Phase 3: the patients will cross over to triamterene or amiloride for 8 weeks. Use the protocol as described in phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Patient with any type of proteinuric kidney diseases
* Aged 18-75
* Proteinuria ≥1g/day
* estimated glomerular filtration rate (eGFR) ≥ 30ml/min/1.73m2

Exclusion Criteria:

* Clinical evidences of lupus nephritis, or HIV associated nephropathy
* eGFR <30ml/min/1.73m2
* Requirement for treatment with mineralocorticoid receptor antagonists (spironolactone, eplerenone)
* Status post kidney transplant
* Received glucocorticoid steroids within six months
* Serum K >4.8 mmol/L
* Total carbon dioxide <17 mmol/L
* Hemoglobin <10 g/dl
* Contraindicated or allergic to loop diuretics or potassium sparing diuretics
* Abnormal liver function tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
24 hr urine protein excretion | 20 weeks
  Identify changes in 24 hr urine protein excretion throughout the 3 phases of the study.

SECONDARY OUTCOMES:
urine plasmin activity | 20 weeks
  examine urine plasmin activity during the 3 phases of the study. Serum and urine plasmin will be measured by gelatin-PAGE zymography.
urine plasminogen activity | 20 weeks
  examine urine plasminogen activity during the 3 phases of the study. urine plasminogen will be measured by gelatin-PAGE zymography.
urine suPAR concentration | 20 weeks
  examine urine suPAR concentration during the 3 phases of the study. suPAR concentration will be measured by ELISA kit.
serum suPAR concentration | 20 weeks
  examine serum suPAR concentration during the 3 phases of the study. suPAR concentration will be measured by ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Shen, MD, PhD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Berhane AM, Weil EJ, Knowler WC, Nelson RG, Hanson RL. Albuminuria and estimated glomerular filtration rate as predictors of diabetic end-stage renal disease and death. Clin J Am Soc Nephrol. 2011 Oct;6(10):2444-51. doi: 10.2215/CJN.00580111. Epub 2011 Aug 18. PMID 21852671
- [Background] Blasi F, Carmeliet P. uPAR: a versatile signalling orchestrator. Nat Rev Mol Cell Biol. 2002 Dec;3(12):932-43. doi: 10.1038/nrm977. PMID 12461559
- [Background] Brown EA, Markandu ND, Roulston JE, Jones BE, Squires M, MacGregor GA. Is the renin-angiotensin-aldosterone system involved in the sodium retention in the nephrotic syndrome? Nephron. 1982;32(2):102-7. doi: 10.1159/000182827. PMID 6757778
- [Background] Brown EA, Markandu ND, Sagnella GA, Jones BE, MacGregor GA. Lack of effect of captopril on the sodium retention of the nephrotic syndrome. Nephron. 1984;37(1):43-8. doi: 10.1159/000183206. PMID 6371561
- [Background] Busch AE, Suessbrich H, Kunzelmann K, Hipper A, Greger R, Waldegger S, Mutschler E, Lindemann B, Lang F. Blockade of epithelial Na+ channels by triamterenes - underlying mechanisms and molecular basis. Pflugers Arch. 1996 Sep;432(5):760-6. doi: 10.1007/s004240050196. PMID 8772124
- [Background] Geers AB, Koomans HA, Roos JC, Boer P, Dorhout Mees EJ. Functional relationships in the nephrotic syndrome. Kidney Int. 1984 Sep;26(3):324-30. doi: 10.1038/ki.1984.176. PMID 6392692
- [Background] Randomised placebo-controlled trial of effect of ramipril on decline in glomerular filtration rate and risk of terminal renal failure in proteinuric, non-diabetic nephropathy. The GISEN Group (Gruppo Italiano di Studi Epidemiologici in Nefrologia). Lancet. 1997 Jun 28;349(9069):1857-63. PMID 9217756
- [Background] Hemmelgarn BR, Manns BJ, Lloyd A, James MT, Klarenbach S, Quinn RR, Wiebe N, Tonelli M; Alberta Kidney Disease Network. Relation between kidney function, proteinuria, and adverse outcomes. JAMA. 2010 Feb 3;303(5):423-9. doi: 10.1001/jama.2010.39. PMID 20124537
- [Background] Iishi H, Tatsuta M, Baba M, Yano H, Uehara H, Nakaizumi A. Suppression by amiloride of bombesin-enhanced peritoneal metastasis of intestinal adenocarcinomas induced by azoxymethane. Int J Cancer. 1995 Nov 27;63(5):716-9. doi: 10.1002/ijc.2910630518. PMID 7591290
- [Background] Kellen JA, Mirakian A, Kolin A. Antimetastatic effect of amiloride in an animal tumour model. Anticancer Res. 1988 Nov-Dec;8(6):1373-6. PMID 3218971
- [Background] Laurens WE, Vanrenterghem YF, Steels PS, Van Damme BJ. A new single nephron model of focal and segmental glomerulosclerosis in the Munich-Wistar rat. Kidney Int. 1994 Jan;45(1):143-9. doi: 10.1038/ki.1994.17. PMID 8127003
- [Background] Lewis EJ, Hunsicker LG, Bain RP, Rohde RD. The effect of angiotensin-converting-enzyme inhibition on diabetic nephropathy. The Collaborative Study Group. N Engl J Med. 1993 Nov 11;329(20):1456-62. doi: 10.1056/NEJM199311113292004. PMID 8413456
- [Background] Madsen CD, Ferraris GM, Andolfo A, Cunningham O, Sidenius N. uPAR-induced cell adhesion and migration: vitronectin provides the key. J Cell Biol. 2007 Jun 4;177(5):927-39. doi: 10.1083/jcb.200612058. PMID 17548516
- [Background] Mathieson PW. Proteinuria and immunity--an overstated relationship? N Engl J Med. 2008 Dec 4;359(23):2492-4. doi: 10.1056/NEJMcibr0806881. No abstract available. PMID 19052132
- [Background] Meltzer JI, Keim HJ, Laragh JH, Sealey JE, Jan KM, Chien S. Nephrotic syndrome: vasoconstriction and hypervolemic types indicated by renin-sodium profiling. Ann Intern Med. 1979 Nov;91(5):688-96. doi: 10.7326/0003-4819-91-5-688. PMID 496101
- [Background] Reiser J, Oh J, Shirato I, Asanuma K, Hug A, Mundel TM, Honey K, Ishidoh K, Kominami E, Kreidberg JA, Tomino Y, Mundel P. Podocyte migration during nephrotic syndrome requires a coordinated interplay between cathepsin L and alpha3 integrin. J Biol Chem. 2004 Aug 13;279(33):34827-32. doi: 10.1074/jbc.M401973200. Epub 2004 Jun 14. PMID 15197181
- [Background] Rennke HG. How does glomerular epithelial cell injury contribute to progressive glomerular damage? Kidney Int Suppl. 1994 Feb;45:S58-63. PMID 8158900
- [Background] Sepehrdad R, Chander PN, Oruene A, Rosenfeld L, Levine S, Stier CT Jr. Amiloride reduces stroke and renalinjury in stroke-prone hypertensive rats. Am J Hypertens. 2003 Apr;16(4):312-8. doi: 10.1016/s0895-7061(03)00006-2. PMID 12670749
- [Background] Thuno M, Macho B, Eugen-Olsen J. suPAR: the molecular crystal ball. Dis Markers. 2009;27(3):157-72. doi: 10.3233/DMA-2009-0657. PMID 19893210
- [Background] Trivedi S, Zeier M, Reiser J. Role of podocytes in lupus nephritis. Nephrol Dial Transplant. 2009 Dec;24(12):3607-12. doi: 10.1093/ndt/gfp427. Epub 2009 Sep 3. No abstract available. PMID 19729466
- [Background] Usberti M, Federico S, Meccariello S, Cianciaruso B, Balletta M, Pecoraro C, Sacca L, Ungaro B, Pisanti N, Andreucci VE. Role of plasma vasopressin in the impairment of water excretion in nephrotic syndrome. Kidney Int. 1984 Feb;25(2):422-9. doi: 10.1038/ki.1984.34. PMID 6727137
- [Background] Vande Walle J, Donckerwolcke R, Boer P, van Isselt HW, Koomans HA, Joles JA. Blood volume, colloid osmotic pressure and F-cell ratio in children with the nephrotic syndrome. Kidney Int. 1996 May;49(5):1471-7. doi: 10.1038/ki.1996.207. No abstract available. PMID 8731116
- [Background] Vande Walle JG, Donckerwolcke RA, Koomans HA. Pathophysiology of edema formation in children with nephrotic syndrome not due to minimal change disease. J Am Soc Nephrol. 1999 Feb;10(2):323-31. doi: 10.1681/ASN.V102323. PMID 10215332
- [Background] Wang Y, Jones CJ, Dang J, Liang X, Olsen JE, Doe WF. Human urokinase receptor expression is inhibited by amiloride and induced by tumor necrosis factor and phorbol ester in colon cancer cells. FEBS Lett. 1994 Oct 17;353(2):138-42. doi: 10.1016/0014-5793(94)01032-3. PMID 7926038
- [Background] Wei C, El Hindi S, Li J, Fornoni A, Goes N, Sageshima J, Maiguel D, Karumanchi SA, Yap HK, Saleem M, Zhang Q, Nikolic B, Chaudhuri A, Daftarian P, Salido E, Torres A, Salifu M, Sarwal MM, Schaefer F, Morath C, Schwenger V, Zeier M, Gupta V, Roth D, Rastaldi MP, Burke G, Ruiz P, Reiser J. Circulating urokinase receptor as a cause of focal segmental glomerulosclerosis. Nat Med. 2011 Jul 31;17(8):952-60. doi: 10.1038/nm.2411. PMID 21804539
- [Background] Wei C, Moller CC, Altintas MM, Li J, Schwarz K, Zacchigna S, Xie L, Henger A, Schmid H, Rastaldi MP, Cowan P, Kretzler M, Parrilla R, Bendayan M, Gupta V, Nikolic B, Kalluri R, Carmeliet P, Mundel P, Reiser J. Modification of kidney barrier function by the urokinase receptor. Nat Med. 2008 Jan;14(1):55-63. doi: 10.1038/nm1696. Epub 2007 Dec 16. PMID 18084301
- [Background] Wei C, Trachtman H, Li J, Dong C, Friedman AL, Gassman JJ, McMahan JL, Radeva M, Heil KM, Trautmann A, Anarat A, Emre S, Ghiggeri GM, Ozaltin F, Haffner D, Gipson DS, Kaskel F, Fischer DC, Schaefer F, Reiser J; PodoNet and FSGS CT Study Consortia. Circulating suPAR in two cohorts of primary FSGS. J Am Soc Nephrol. 2012 Dec;23(12):2051-9. doi: 10.1681/ASN.2012030302. Epub 2012 Nov 8. PMID 23138488
- [Background] Wei Y, Waltz DA, Rao N, Drummond RJ, Rosenberg S, Chapman HA. Identification of the urokinase receptor as an adhesion receptor for vitronectin. J Biol Chem. 1994 Dec 23;269(51):32380-8. PMID 7528215
- [Background] Wu S, Murrell GA, Wang Y. Interferon-alpha (Intron A) upregulates urokinase-type plasminogen activator receptor gene expression. Cancer Immunol Immunother. 2002 Jul;51(5):248-54. doi: 10.1007/s00262-002-0275-5. Epub 2002 Apr 9. PMID 12070711
- [Background] Zhang B, Xie S, Shi W, Yang Y. Amiloride off-target effect inhibits podocyte urokinase receptor expression and reduces proteinuria. Nephrol Dial Transplant. 2012 May;27(5):1746-55. doi: 10.1093/ndt/gfr612. Epub 2011 Nov 9. PMID 22076430
- [Derived] Shen W, Alshehri M, Desale S, Wilcox C. The Effect of Amiloride on Proteinuria in Patients with Proteinuric Kidney Disease. Am J Nephrol. 2021;52(5):368-377. doi: 10.1159/000515809. Epub 2021 May 6. PMID 33957621